CLINICAL TRIAL: NCT04327518
Title: Clinical Investigation of Rotational Stability of the TECNIS® Toric II Intraocular Lens
Brief Title: Evaluation of the Rotational Stability of the Tecnis Toric II IOL
Acronym: STEELE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NXGT-202-QROS
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Results first posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Cataract; Corneal Astigmatism
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- TECNIS® Toric II (Experimental): Subjects will be implanted in one or both eyes with the study lens
  Interventions: Device: TECNIS® Toric II

INTERVENTIONS:
Device: TECNIS® Toric II — Toric Intraocular Lens

SUMMARY:
This is a prospective, multicenter, single-arm, open-label clinical study of the commercially available TECNIS Toric II IOL. The study will be conducted in up to 192 subjects needing unilateral or bilateral cataract surgery in up to 8 sites in United States (US). The subjects will be followed for up to 3-months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum 22 years of age;
2. Unilateral or Bilateral cataracts for which cataract extraction and posterior chamber IOL implantation have been planned;
3. Pre-existing corneal astigmatism of one diopter or greater;
4. Predicted residual refractive cylinder based on toric IOL calculator, considering surgically induced astigmatism (SIA) and posterior corneal astigmatism (PCA) must be ≤0.50 D;
5. Potential for postoperative BCDVA of 20/30 Snellen or better;
6. Clear intraocular media other than cataract in each eye;
7. Availability, willingness and sufficient cognitive awareness to comply with examination procedures and study visits;
8. Signed informed consent form (ICF) and health insurance portability and accountability act (HIPAA) authorization;
9. Ability to understand and respond to a questionnaire in English.

Exclusion Criteria:

1. Irregular corneal astigmatism;
2. Any corneal pathology/abnormality other than regular corneal astigmatism or corneal instability due to contact lens wear;
3. Previous corneal or intraocular surgery;
4. Inability to focus or fixate for prolonged periods of time (e.g., due to strabismus, nystagmus, etc.);
5. Any pupil abnormalities (non-reactive, fixed, or abnormally shaped pupils);
6. Dilated pupil size of < 6.0 mm;
7. Recurrent severe anterior or posterior segment inflammation or uveitis;
8. Subjects with conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration, including pseudoexfoliation, trauma, or posterior capsule defects;
9. Known ocular or systemic disease that, in the opinion of the investigator, may affect visual acuity or require surgical intervention during the course of the study, [macular degeneration, cystoid macular edema, proliferative diabetic retinopathy (severe), uncontrolled glaucoma, irregular corneal astigmatism, choroidal hemorrhage, concomitant severe eye disease, extremely shallow anterior chamber, microphthalmos, non-age related cataract, severe corneal dystrophy, severe optic nerve atrophy, etc.];
10. Use of systemic or ocular medications (e.g., Flomax) that may affect vision including prior, current, or anticipated use during the course of the study that may, in the opinion of the investigator, confound the outcome or increase the risk to the subject (e.g., poor dilation or a lack of adequate iris structure to perform standard cataract surgery);
11. Patient is pregnant, plans to become pregnant, is lactating or has another condition associated with the fluctuation of hormones that could lead to refractive changes;
12. Concurrent participation or participation within 30 days prior to the preoperative visit in any other clinical study.
13. Planned monovision correction (eye designated for near correction)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision Clinical Trials, Study Director — Johnson & Johnson Surgical Vision
Locations (7):
- United States (7):
  - Empire Eye and Laser Center, Inc., Bakersfield, California
  - University of California, Los Angeles, California
  - Jones Eye Clinic, Sioux City, Iowa
  - Vance Thompson Vision, ND, West Fargo, North Dakota
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - JW Eye Associates, P.A. DBA Key-Whitman Eye Center, Dallas, Texas
  - Texas Eye & Laser Center, P.A., Hurst, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 125 subjects were enrolled. A total of 202 eyes were implanted with the TECNIS Toric II IOL in at least one eye: 80 subjects were treated bilaterally (77 subjects with study lens on both eyes, 3 subjects with non-study lens on first eye and study lens on second eye) and 45 subjects were treated unilaterally. All implanted subjects were examined through 3-months postoperatively.
Units Other Than Participants: Eyes
Groups:
- Tecnis Toric II IOl: Study Lens
Period: Overall Study
Arm/Group | Tecnis Toric II IOl
Started | 125; 202 Eyes
Completed | 124; 200 Eyes
Not Completed | 1; 2 Eyes

BASELINE CHARACTERISTICS:
Arm/Group | Tecnis Toric II IOL
Number analyzed (Participants) | 125
Age, Customized [Number; unit: Participants]
  <60 years | 17
  60-69 years | 47
  70-79 years | 53
  >+80 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 118
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 112
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With ≤ 5º Lens Axis Misalignment From the Intended IOL Axis of Orientation at the 1-week Postoperative Visit
Description: Absolute difference between intended IOL axis of orientation (immediately at the end of surgery) and follow-up visit(s) were measured by a photographic based method.
Time Frame: 1 week postoperative
Population: All Toric II Eyes with Valid Axis Data
Measure: Number (95% Confidence Interval); unit: Percentage of Eyes
Units Other Than Participants: Eyes
Arm/Group | Tecnis Toric II IOL
Number analyzed (Participants) | 119
Number analyzed (Eyes) | 191
Percentage of Eyes | 99.5 [98.5 to 100]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Tecnis Toric II IOL
All-Cause Mortality (participants affected / at risk) | 0/125
Serious Adverse Events (participants affected / at risk) | 4/125
Other Adverse Events (participants affected / at risk) | 0/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tecnis Toric II IOL (N=125)
Myocardial Infarction (Cardiac disorders) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1)
Cystoid Macular Edema (Eye disorders) | 1 (1)
Pulmonary Bilateral embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyphema (Eye disorders) | 1 (1)
Hemorrhagic Choroidal Detachment (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review results communication prior to public release and can embargo communications regarding trial results at anytime.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT04327518/Prot_SAP_001.pdf